CLINICAL TRIAL: NCT03231852
Title: Patient Perceptions and Willingness to Enroll in Clinical Trials
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Linda R Duska, Professor, Department of Obstetrics and Gynecology, University of Virginia
Other Study IDs: 19844
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Cancer, Clinical Trials
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: Women with a gynecologic malignancy will complete several surveys to assess their willingness to participate in clinical trials.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Attitudes and Randomized Trial Questionnaire (ARTQ), Hospital Anxiety and Depression Scale, Perception Survey

SUMMARY:
The objective of our study is to determine which factors affect willingness to participate in gynecologic oncology clinical trials. Women with a diagnosis of gynecologic malignancy will be approached to complete a survey assessing willingness to participate in clinical trials. The validated Attitudes and Randomized Trials Questionnaire (ARTQ) will be used to assess willingness to participate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gynecologic malignancy
* English or Spanish literate

Exclusion Criteria:

* Prior enrollment in a clinical trial
* Currently pregnant
* Currently incarcerated

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All women presenting to the gynecologic oncology clinic meeting the inclusion/exclusion criteria will be approached to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Willingness to Participate in Clinical Trials | 6 months
  Bivariate outcome derived from ARTQ survey

CONTACTS AND LOCATIONS:
Overall Officials: Linda Duska, MD, MPH, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No